CLINICAL TRIAL: NCT01101984
Title: A Randomized, Parallel- Group Comparison Study of DE-089 Ophthalmic Solution in Patients With Dry Eye (Comparison With 0.1% Sodium Hyaluronate Ophthalmic Solution) - A Multinational Study -
Brief Title: Study of DE-089 Ophthalmic Solution in Patients With Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08901
Record Dates: First submitted 2010-04-07; First posted 2010-04-12 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- DE-089 (Experimental): DE-089 ophthalmic solution
  Interventions: Drug: diquafosol ophthalmic solution; Drug: 0.1% sodium hyaluronate ophthalmic solution.
- HA (Active Comparator): 0.1% sodium hyaluronate ophthalmic solution
  Interventions: Drug: 0.1% sodium hyaluronate ophthalmic solution.

INTERVENTIONS:
Drug: diquafosol ophthalmic solution — DE-089 topical ocular application, 6 times daily for 4 weeks.
  Other Names: HA
  Arms: DE-089
Drug: 0.1% sodium hyaluronate ophthalmic solution. — 0.1% HA topical ocular application, 6 times daily for 4 weeks.

SUMMARY:
Safety and efficacy of DE-089 ophthalmic solution in patients with dry eye will be evaluated in comparison with sodium hyaluronate ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

* Those who show:

  * Keratoconjunctival disorder confirmed with vital dye staining
  * Abnormal Schirmer score results

Exclusion Criteria:

* Eye disease that needs therapy other than that for dry eye
* Those who need to wear contact lenses during the clinical study

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-02; Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Changes in the fluorescein and rose bengal staining score | 2 weeks and 4 weeks from baseline.
  1. Changes in the fluorescein staining score at Week 4 / at the time of discontinuation (non-inferiority)
  2. Changes in the rose bengal staining score at Week 4 / at the time of discontinuation (superiority)

SECONDARY OUTCOMES:
Changes in tear film breakup time (second) | 2 weeks and 4 weeks from baseline.
  Changes in tear film breakup time (second) 2 weeks, 4 week after the study / at the discontinuation

CONTACTS AND LOCATIONS:
Locations (2):
- Eye & Ear Hospital of Fudan University, Shanghai, China
- Singapore Eye Research Institute, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Gong L, Sun X, Ma Z, Wang Q, Xu X, Chen X, Shao Y, Yao K, Tang L, Gu Y, Yuan H, Chua WH, Chuan JC, Tong L. A randomised, parallel-group comparison study of diquafosol ophthalmic solution in patients with dry eye in China and Singapore. Br J Ophthalmol. 2015 Jul;99(7):903-8. doi: 10.1136/bjophthalmol-2014-306084. Epub 2015 Jan 28. PMID 25631485